CLINICAL TRIAL: NCT01393821
Title: A Randomized, Double-Blind Placebo-Controlled Exploration of a Topical Menadione-Containing Lotion to the Face for Prevention and Palliation of Epidermal Growth Factor Receptor Inhibitor-Induced Cutaneous Discomfort and Psychological Distress
Brief Title: Menadione Topical Lotion in Treating Skin Discomfort and Psychological Distress in Patients With Cancer Receiving Panitumumab, Erlotinib Hydrochloride, or Cetuximab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC10C9; NCI-2011-01047 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11-001566 (Other: Mayo Clinic Institutional Review Board); R21CA134432 (NIH)
Record Dates: First submitted 2011-06-27; First posted 2011-07-13 (Estimated); Results first posted 2019-10-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Dermatologic Complications; Malignant Neoplasm; Pain
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (lotion) (Experimental): Patients apply menadione topical lotion BID for 28 days.
  Interventions: Drug: menadione topical lotion; Other: questionnaire administration; Procedure: management of therapy complications
- Arm II (placebo) (Placebo Comparator): Patients apply topical placebo lotion BID for 28 days.
  Interventions: Other: placebo; Other: questionnaire administration

INTERVENTIONS:
Drug: menadione topical lotion — Given topically
  Arms: Arm I (lotion)
Other: placebo — Given topically
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: questionnaire administration — Ancillary studies
Procedure: management of therapy complications — Given menadione topical lotion
  Other Names: complications of therapy, management of
  Arms: Arm I (lotion)

SUMMARY:
This clinical trial studies menadione topical lotion in treating skin discomfort and psychological distress in patients with cancer receiving panitumumab, erlotinib hydrochloride, or cetuximab. Menadione topical lotion may prevent rash or other skin discomfort and help alleviate psychological distress and pain in patients receiving treatment with panitumumab, erlotinib hydrochloride, or cetuximab

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Explore the effectiveness of a menadione topical lotion to the face to prevent cutaneous and psychological discomfort from epidermal growth factor receptor (EGFR) inhibitors.

SECONDARY OBJECTIVES:

I. Explore the adverse event profile of a menadione topical lotion to the face to prevent rash from EGFR inhibitors.

II. Explore whether rash or adverse events worsen over a 4 week period after this 4-week intervention.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients apply menadione topical lotion twice daily (BID) for 28 days.

ARM II: Patients apply topical placebo lotion BID for 28 days.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Patient scheduled to start an epidermal growth factor receptor inhibitor (must be one of these three: panitumumab, erlotinib, cetuximab) within the next 3 days or patient has already started the epidermal growth factor receptor inhibitor but has not been on it for longer than 3 days and has no signs or symptoms potentially suggestive of EGFR inhibitor toxicity.
* Ability to reliably apply Menadione Topical Lotion / placebo twice a day to the face.
* Ability to complete questionnaire(s) by themselves or with assistance.
* Negative pregnancy test (serum or urine) done ≤ 7 days prior to registration, for women of childbearing potential only.
* Willing to have photographs taken to assess rash.

Exclusion Criteria:

* Any active facial and/or chest rash, including adult acne, at the time of randomization.
* Cutaneous metastases, skin cancer, or a history of precancerous skin lesions involving the face and/or chest.
* Use of topical corticosteroids on the face and/or chest at the time of study entry or their anticipated use in the next 8 weeks.
* Any type of ongoing therapy for rash.
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception since this study involves agents that have known genotoxic, mutagenic and teratogenic effects
* Use of any antibiotic at the time of study or their anticipated use in the 8 weeks immediately following study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-01-23 (Actual); Primary Completion 2013-05-11 (Actual); Study Completion 2018-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, M.D., Study Chair — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Campus in Arizona, Phoenix, Arizona
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Menadione): Patients apply menadione topical lotion BID for 28 days.
- Arm B (Placebo): Patients apply topical placebo lotion BID for 28 days.
Period: Overall Study
Arm/Group | Arm A (Menadione) | Arm B (Placebo)
Started (eligible participants) | 14 | 13
Completed (evaluable for primary endpoint) | 9 | 10
Not Completed | 5 | 3
Not completed — Cancel | 1 | 1
Not completed — not evaluable for primary endpoint | 4 | 2

BASELINE CHARACTERISTICS:
Population: Excludes cancel patients who never received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Menadione) | Arm B (Placebo) | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.3) | 64.3 (12.6) | 63.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 7 | 6 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 Face Pain Score Measuring Cutaneous Discomfort
Description: Change from baseline to Week 4 Face pain score measuring cutaneous discomfort. Face pain scale question ("How would you describe how your face feels?") with a 0-10 Face Pain Scale, where 0 = No pain/burning and 10 = worst possible pain/burning.
Time Frame: From Baseline to Week 4
Population: Patients who completed the face pain question at baseline and week 4 are included in this analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm A (Menadione) | Arm B (Placebo)
Number analyzed (Participants) | 8 | 10
score on a scale | 2.0 [0.0 to 4.0] | 3.0 [0.0 to 5.0]
Statistical Analysis 1: Comparison: Arm A (Menadione) vs Arm B (Placebo); Test type: Superiority; p = 0.6311, Kruskal-Wallis

2. Secondary Outcome: The Number of Patients Experiencing Worst Toxicity
Description: The number of patients experiencing treatment-related adverse events (toxicities) is reported below. The maximum grade toxicity (worst toxicity) is reported by arm.
Time Frame: Up to 8 weeks
Population: Excludes cancel patients who never received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Menadione) | Arm B (Placebo)
Number analyzed (Participants) | 13 | 12
Participants
  Grade 1 | 3 | 3
  Grade 2 | 7 | 6
  Grade 3 | 3 | 3

3. Secondary Outcome: Long-term Cutaneous Discomfort as Measured by the Change From Baseline in Face Pain Scale at 4 Weeks (Treatment-regimen Estimand)
Description: Least Squares mean (LS) of the Face Pain Scale change from baseline at week 4 was adjusted by treatment, week, race, gender, age (<=50 years/>50 years), and EGFR, via a MMRM analysis. Face pain scale question ("How would you describe how your face feels?") with a 0-10 Face Pain Scale, where 0 = No pain/burning and 10 = worst possible pain/burning.
Time Frame: Baseline, 4 weeks
Population: Excludes cancel patients who never received treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Arm A (Menadione) | Arm B (Placebo)
Number analyzed (Participants) | 13 | 12
score on a scale | 2.1820 (0.5003) | 1.8244 (0.4376)

4. Secondary Outcome: Long-term Psychosocial Discomfort as Measured by the Change From Baseline in Psychological Distress Score at 4 Weeks (Treatment-regimen Estimand)
Description: Least Squares mean (LS) of the Psychological Distress Score change from baseline at week 4 was adjusted by treatment, week, race, gender, age (<=50 years/>50 years), and EGFR, via a MMRM analysis. Psychological Distress question ("How often have you been bothered by embarrassment about your face?") with a 0-6 scale, where 0 = Never bothered and 6 = Always bothered.
Time Frame: Baseline, Week 4
Population: Excludes cancel patients who never received treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Arm A (Menadione) | Arm B (Placebo)
Number analyzed (Participants) | 13 | 12
score on a scale | 0.7196 (0.3436) | 1.1891 (0.3043)

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Description: Excludes cancel patients who never received treatment.
Arm/Group | Arm A (Menadione) | Arm B (Placebo)
All-Cause Mortality (participants affected / at risk) | 2/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/12 | 1/13
Other Adverse Events (participants affected / at risk) | 11/12 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Menadione) (N=12) | Arm B (Placebo) (N=13)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Menadione) (N=12) | Arm B (Placebo) (N=13)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (2) | 1 (1)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6) | 9 (11)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (16) | 12 (16)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes